CLINICAL TRIAL: NCT05337657
Title: A Multicenter, Open-label, Phase Ib Clinical Trial of GB491 in Combination With Letrozole in Previously Untreated Patients With HR-positive, HER2-negative Advanced Breast Cancer
Brief Title: A Phase Ib Study of GB491 Plus Letrozole in Patients With Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Genor Biopharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GB491-005
Record Dates: First submitted 2021-12-21; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2021-12

CONDITIONS: Advanced Breast Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- GB491+Letrozole (Experimental)
  Interventions: Drug: GB491+Letrozole

INTERVENTIONS:
Drug: GB491+Letrozole — Drug：The dose of GB491 is 150 mg, which should be taken with a meal and taken twice daily at approximately the same time each day, approximately 12 hours apart

SUMMARY:
GB491-005 is a multicenter, open-label, phase Ib Clinical Trial study to evaluate the safety, pharmacokinetic (PK), pharmacodynamic (PD) activity, and preliminary anti-tumor activity of GB491 in combination with Letrozole in Previously Untreated Patients with HR-positive, HER2-negative Advanced Breast Cancer

ELIGIBILITY:
Inclusion Criteria:

1. Females of 18 years of age or older at study screening
2. Histologically or cytologically confirmed locally advanced or advanced metastatic breast cancer that is not amenable to curative surgical resection or radiation therapy
3. The subject has been diagnosed with ER-positive breast cancer in the local laboratory
4. The subject has HER2-negative breast cancer in the local laboratory
5. Menopausal status is not limited (including Premenopausal/perimenopausal/postmenopausal state)
6. No previous systemic anti-tumor treatment for locally advanced or metastatic breast cancer;
7. According to RECIST V1.1, the patient has at least one measurable lesion that has not been irradiated by radiotherapy and can be evaluated by CT/MRI; If only bone metastases are present, there must be at least one osteolytic bone lesion that can be evaluated by CT/MRI
8. ECOG performance status of 0 or 1
9. Adequate organ and marrow function.
10. The subject of childbearing potential must use one highly effective birth control method from the total duration of the study and 6 months after the last dose of study intervention.
11. Provide informed consent

Exclusion Criteria:

1. Previous treatment with CDK4/6 inhibitors
2. Subjects with known hypersensitivity to any component of GB491 or Letrozole
3. Patients with disease progression or recurrence during or within 1 year after completion of previous endocrine neoadjuvant or adjuvant therapy
4. Known active, uncontrolled, or symptomatic central nervous system metastasis, carcinomatous meningitis, or clinically manifested leptomeningeal disease, cerebral edema, spinal compression or/and tumor progressive growth
5. Visceral crisis
6. Patients with skin lesion only and radiographically non-measurable at baseline
7. Persistent toxicities (CTCAE Grade ≥ 2) caused by previous anticancer therapy, excluding alopecia
8. Major surgical procedure within 4 weeks of the first dose of study treatment or an anticipated need for major surgery, chemotherapy, radiotherapy, any other investigational drug or other anti-cancer therapy during the study
9. Patients who have been on bisphosphonates and denosumab therapy at a stable dose for less than 14 days prior to randomization
10. Patients who have received limited field radiotherapy in 2 weeks or extended field radiotherapy in 4 weeks before randomization or radiation with more than 30% of the bone marrow
11. Subjects use drugs or fruits containing strong inducers or inhibitors of CYP3A4/5, or drugs with narrow therapeutic window that are mainly metabolized by CYP3A4/5 in 14 days before randomization
12. Patients with long-term systematic use of corticosteroids
13. Any severe and/or uncontrollable medical conditions
14. Patients with severely impaired lung function
15. Known history of HIV infection or history of HIV seropositivity
16. Resting QTcF > 480 msec or there is a medical history of QTcF prolongation
17. Subjects have significant hepatic disease
18. Coagulation abnormalities
19. Refractory nausea and vomiting, inability to swallow the formulated product, or other disease or clinical status would preclude adequate absorption, distribution, metabolism, or excretion of GB491
20. Previous allogeneic bone marrow transplant
21. Inflammatory breast cancer;
22. Subjects with a history of other primary malignancies, except for non-melanoma skin cancer and cervical cancer in situ disease-free status ≥ 3 years
23. Lactating women
24. Unlikely to comply with study procedures, restrictions, and requirements
25. Judgment by the investigator that the patient should not participate into the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-12-12 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
DLT | During Cycle 1 (up to 28 days)
  Number of Participants with Dose-Limiting Toxicities for GB491 in Combination with Letrozole
AE | From Baseline until 30 days after the last treatment
  Number of Participants with Adverse Events by Severity, According to National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 (NCI-CTCAE v5.0)

SECONDARY OUTCOMES:
PFS | Approximately 2 years
  To assess the progression free survival assessed by investigator
ORR | Approximately 2 years
  To assess the objective response rate for GB491 in Combination with Letrozole
DOR | Approximately 2 years
  To assess the duration of response for GB491 in Combination with Letrozole
DCR | Approximately 2 years
  To assess the disease control rate for GB491 in Combination with Letrozole
CBR | Approximately 2 years
  To assess the clinical benefit rate for GB491 in Combination with Letrozole by investigator
Plasma Concentration of GB491 | At predefined intervals from Cycle 1, Day 1 & Day 15; Cycle 2, Day 1 (each cycle is 28 days)
  Plasma Concentration of GB491 Over Time
Plasma Concentration of Letrozole | At predefined intervals from Cycle 1, Day 1 & Day 15; Cycle 2, Day 1 (each cycle is 28 days)
  Plasma Concentration of Letrozole Over Time

CONTACTS AND LOCATIONS:
Overall Officials: Xichun Hu, PhD, Principal Investigator — Fudan University; Jian Zhang, PhD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China